CLINICAL TRIAL: NCT02699138
Title: Obstructive Sleep Apnea and Arousal Threshold in Patients With Post-traumatic
Brief Title: Obstructive Sleep Apnea and Arousal Threshold in Patients With Post-traumatic Stress Disorder
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Research fellow left institution
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert L. Owens, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UCSD151424
Record Dates: First submitted 2016-02-24; First posted 2016-03-04 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Sleep Apnea, Obstructive; Post-Traumatic Stress Disorders
MeSH Terms: conditions — Sleep Apnea Syndromes; Stress Disorders, Post-Traumatic | interventions — Trazodone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Trazodone (Experimental): To determine effect of trazodone on quality of sleep as measured by apnea hypopnea index in subjects with obstructive sleep apnea and PTSD on routine overnight polysomnogram.
  Interventions: Drug: Trazodone; Device: Epiglottic catheter
- Placebo (Placebo Comparator): To compare placebo outcomes against administration of trazodone
  Interventions: Drug: Placebo; Device: Epiglottic catheter

INTERVENTIONS:
Drug: Trazodone — 100mg of trazodone to be administered orally once.
  Arms: Trazodone
Drug: Placebo — Compounded sugar pill
  Arms: Placebo
Device: Epiglottic catheter — Catheter that can be placed through the nose to a position behind the tongue to monitor for upper airway obstruction and to measure changes in pressure below the obstruction.

SUMMARY:
Obstructive sleep apnea (OSA) has traditionally been attributed only to a collapsible upper airway. However, it is increasingly recognized that multiple additional non-anatomical mechanisms contribute to the disease. Higher rates of OSA in patients with post-traumatic stress disorder (PTSD) than in those without PTSD have been reported however the mechanism behind this increased prevalence has not been investigated. Our hypothesis is that patients with PTSD have a predisposition to OSA due to a lower respiratory arousal threshold (wake up too easily) than patients without PTSD. The goal of this project will be to study and compare the ArTH in patients with PTSD and those without. In addition, we plan to see whether medications can be used to increase the arousal threshold and treat OSA in patients with PTSD.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a clinically relevant disease that is associated with cardiovascular, metabolic, and neurocognitive consequences. OSA is a very common disease; the Wisconsin Sleep Cohort Study found that OSA affects 2% of women and 4% of men aged 30-60. However, these data predate the obesity epidemic and use of more modern diagnostic equipment, such that more recent studies have reported prevalences of moderate to severe OSA as high as 24% in women and 49% in men.

The prevalence of OSA has been found to be particularly high in patients suffering from post-traumatic stress disorder (PTSD). One study of veterans with combat related PTSD found that 67.3% of this population was diagnosed with OSA after undergoing polysomnography. This finding is consistent with those of Mysliwiec et al who found rates of OSA in 63% of post-deployment soldiers and 51% of active duty soldiers. Despite increased recognition of this association, there has been little progress in establishing a pathophysiological link between the two diseases, and no study to our knowledge examining the possibility that PTSD might drive the development of OSA. Furthermore, individuals with PTSD have been found to have significantly lower compliance with continuous positive airway pressure (CPAP) therapy than the general population, with claustrophobia, mask discomfort, and air hunger as the most commonly cited reasons for non-adherence. Despite this, studies have shown both benefit in sleep quality and PTSD related nightmares with OSA treatment. Alternative OSA therapies are therefore particularly important in this group, but will rely on determination of targets other than those treated by CPAP.

While a propensity towards upper airway collapse, as seen in obesity, has classically been considered the principle determinate of OSA pathogenesis, more recent work has shown that non-anatomical variables including the ventilatory arousal threshold (ArTH) are also important. During wakefulness pharyngeal dilator muscles remain active to maintain airway patency however during sleep these muscles lose activity in all individuals but in those with OSA airway collapse occurs and results hypoxia and hypercapnia. Both accumulation of carbon dioxide and increased negative pressure can cause recruitment of the upper airway dilator muscles resulting in pharyngeal patency if sleep is maintained. Cortical arousal during apnea for most individuals represents a protective mechanism as the airway is restored with resolution of hypoxia and hypercarbia. However individuals with low ArTH (individuals who wake easily) do not have sufficient time for accumulation of respiratory stimuli, recruitment of pharyngeal muscles is then unable to occur which results in disruption of sleep. ArTH is variable amongst individuals and is dependent on the magnitude of negative intrathoracic pressure tolerated before awakening occurs and is independent from other factors.

A central feature of PTSD is a state of persistent hyperarousal that chronically persists following a traumatic event. Individuals with PTSD have been found to have important physiologic changes of the hypothalamic-pituitary axis (HPA) and sympathoadrenal system including increased levels of sympathetic neurotransmitters such as norepinephrine and increased activity of α2-adrenergic and glucocortocoid receptors. Both the HPA and sympathetic nervous system are associated with attention and arousal. Prolonged activation of these systems has been shown to induce important biochemical changes associated with disordered sleep. Indeed, studies in norepinephrine deficient knockout mice have demonstrated that increased stimulus is required to induce cortical arousal in the norepinephrine deficient mice and results in higher acoustic ArTH when compared to controls. Our hypothesis is that patients suffering from PTSD will have a lower ArTH when compared to subjects without PTSD. This work is significant because if lower ArTH is associated with PTSD these patients may benefit from therapies that raise the ArTH.

Prior studies have indicated that trazodone, a serotonin reuptake inhibitor commonly used for insomnia and occasionally for depression, may raise the arousal threshold without suppressing upper airway muscle activity. This medication therefore presents a potentially attractive alternative treatment to CPAP therapy for patients with OSA related to a low arousal threshold.

ELIGIBILITY:
Inclusion Criteria:

* Normal sleep study aside from elevated AHI
* Prior home sleep test (HST) or polysomnogram with results consistent with mild, moderate, or severe sleep apnea. If a sleep study has not been performed in the past, the participant will be offered an HST and included if OSA is confirmed on HST.
* PTSD as diagnosed by psychiatrist, psychologist, or other licensed mental health professional

Exclusion Criteria:

* Any known cardiac (apart from treated hypertension), symptomatic pulmonary (including asthma), renal, neurologic (including epilepsy), neuromuscular, or hepatic disease.
* Pregnant women.
* History of hypersensitivity to Afrin, Lidocaine, or Trazodone
* History of bleeding diathesis and/or gastrointestinal bleeding.
* Daily use of any sedative medications that may affect sleep or breathing, including benzodiazepines, opioids, or hypnotics.
* A psychiatric disorder, other than mild depression or PTSD; e.g. schizophrenia, bipolar disorder, major depression, panic or anxiety disorders.
* Substantial cigarette (>5/day), alcohol (>3oz/day) or use of illicit drugs.
* More than 10 cups of beverages with caffeine (coffee, tea, soda/pop) per day.
* Subjects with oxyhemoglobin desaturations to <70% on the initial PSG (Aim 1) will be excluded from participation in Aim 2.
* Current, everyday use of continuous positive airway pressure therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Respiratory arousal threshold | 8 hours
  Arousal threshold will be measured by epiglottic catheter placement during routine polysomnograph. Respiratory arousal threshold is measured by standard criteria and determined by difference in the terminal pressure measured prior to cortical arousal on EEG and the baseline epiglottic pressure.
Apnea hypopnea index | 8 hours
  Severity of obstructive sleep apnea measured by the apnea hypopnea index. Measured by standard sleep scoring criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Owens, MD, Principal Investigator — UCSD
Locations (1):
- University of California San Diego, San Diego, California, United States